CLINICAL TRIAL: NCT00515983
Title: Phase I Clinical Trial of a Therapeutic Vaccine Composed of Autologous Dendritic Cells Loaded With Allogeneic Apoptotic Tumor Cells in Patients With Melanoma Stages IIB, IIC, III and IV
Brief Title: Vaccination of Melanoma Patients With Dendritic Cells Loaded With Allogeneic Apoptotic-Necrotic Melanoma Cells
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: José Mordoh, M.D., Ph.D. (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 4484/04
Record Dates: First submitted 2007-08-10; First posted 2007-08-14 (Estimated); Last update posted 2007-08-14 (Estimated); Status verified 2007-08

CONDITIONS: Melanoma
Keywords: melanoma; dendritic cells; apoptotic/necrotic cells; therapeutic vaccine
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Who Masked: Participant

INTERVENTIONS:
Biological: DC/Apo-Nec

SUMMARY:
Background: Sixteen melanoma patients (1 stage IIC, 8 stage III, and 7 stage IV) were treated in a Phase I study to evaluate safety and immune responses, with a vaccine (DC/Apo-Nec) composed of autologous dendritic cells (DCs) loaded with a mixture of apoptotic/necrotic melanoma cell lines (Apo-Nec).

Methods: PBMC were obtained from leukapheresis and DCs were generated from monocytes cultured in the presence of GM-CSF and IL-4 in serum-free medium. Immature DCs (iDCs) were loaded with gamma-irradiated Apo-Nec cells and injected id without adjuvant. Cohorts of four patients were given four vaccines with 5, 10, 15, or 20 x106 DC/Apo-Nec per vaccine, two weeks apart.

Results: The vaccine was well tolerated in all patients. Toxicity to vaccine was mild, and the toxicity-limiting dose has not been reached. We found that 42.3 ±13.7 % melanoma patients´ iDCs were able to phagocyte Apo-Nec cells wich induced DCs maturation, as evidenced by increased expression of CD83, CD80, CD86, HLA class I and II compared to iDCs. Also, after phagocytosis, a 75.2 ±16 % reduction in Dextran-FITC endocytosis was observed compared to iDCs. CCR7 was upregulated upon Apo-Nec phagocytosis in DCs from all patients and accordingly in vitro DC/Apo-Nec cells were able to migrate towards MIP-3 beta. The DTH score increased significatively in the patients after the first vaccination and slightly decreased by the fourth vaccine (Mann-Whitney Test, p<0.05). For patient #1 a positive DTH reaction was detected to her own tumor irradiated cells. The presence of CD8+ T lymphocytes specific to gp100 and Melan A/MART-1 Ags were studied by tetramers binding in HLA-A*0201 patients (7 /15 patients) before and after vaccination. Two patients who remain NED increased Ags their specific T lymphocytes after vaccination. No humoral responses to Apo-Nec cells were detected. With a mean follow-up of 44.5 months post-surgery, the stage IIC pt is NED, 7/8 stage III pts are NED and 7/7 stage IV patients have progressed.

Conclussions: We conclude that DC/Apo-Nec vaccine is well tolerated, it induces specific immunity against melanoma Ags and in stage III patients it may prolong disease-free survival, affording protection from relapse in an adjuvant setting.

ELIGIBILITY:
Inclusion Criteria:

* histologically confirmed cutaneous melanoma stages IIB, IIC, III or IV (AJCC)
* pts with minimal or non-detectable disease (NED) after surgery as asserted by CAT scans. Melanoma pts with unknown primary tumor site could be included in the study
* life expectancy > 6 months
* ages:from 15 to 60 years
* performance status (ECOG) 0 or 1
* pts with stage III disease had to be previously treated with IFN-alpha, and either finished the treatment or suspended it due to disease progression, toxicity or other clinical reasons. Alternatively, those pts who had not started IFN-alpha within six months after surgery could be included in this study
* a suitable venous access for the leukapheresis procedure
* laboratory eligibility criteria included: hemoglobin > 10 gr %; WBC count > 4800/mm3, platelets > 150.000/mm3, total and direct bilirubin, serum oxalacetic transaminase and glutamic pyruvic transaminase < 1.5 fold the upper normal value; LDH < 450 mU/ml
* absence of pregnancy, with serum βHCG determined one week before vaccination in premenopausal women
* serum creatinine < 1.4 mg %
* no chemotherapy, radiotherapy or any biological treatments during the previous month
* no concurrent medication with corticosteroids or NSAIDs
* l no active brain metastases m- normal ECG
* all pts gave written informed consent before inclusion in the Study.

Exclusion Criteria:

* Ocular melanoma or melanoma of mucosa
* Active brain metastases
* Other previous carcinoma (with the exeption of cervical or in situ basal cells carcinoma adequately treated)
* Pregnant or breast-feeding women
* Cardiac Arythmia, severe heart disease.
* Bacterial, mycotic or viral serious infections ( > grade 2 according to NCI common toxicity criteria)
* HIV, B or C Hepatitis previous infection
* Primary or secondary immunodeficiencies
* Other diseases that require treatment with regular corticoids or non steroids anti-inflammatory drugs or COX-2 inhibitors

Ages: 17 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2004-10; Study Completion 2005-12 (Actual)

PRIMARY OUTCOMES:
Toxicity measured according to the NCI-Common Toxicity Criteria. | 115 days follow up per Subject (Trial duration)
Induction of immune responses associated to different vaccine doses | 115 days follow up per subject (Trial duration)

SECONDARY OUTCOMES:
Feasibility | 115 days follow up per subject (Trial duration)

CONTACTS AND LOCATIONS:
Overall Officials: José Mordoh, MD,PhD, Study Director
Locations (1):
- Instituto Médico Alexander Fleming, Buenos Aires, Buenos Aires F.D., Argentina

REFERENCES:
- [Derived] von Euw EM, Barrio MM, Furman D, Levy EM, Bianchini M, Peguillet I, Lantz O, Vellice A, Kohan A, Chacon M, Yee C, Wainstok R, Mordoh J. A phase I clinical study of vaccination of melanoma patients with dendritic cells loaded with allogeneic apoptotic/necrotic melanoma cells. Analysis of toxicity and immune response to the vaccine and of IL-10 -1082 promoter genotype as predictor of disease progression. J Transl Med. 2008 Jan 25;6:6. doi: 10.1186/1479-5876-6-6. PMID 18221542